CLINICAL TRIAL: NCT00440856
Title: Reduction in Leg and Back Pain Following Lumbar Microdiscetomy in Those Shown the Removed Disc Fragments After the Operation: a Double Blind Randomized Control Trial.
Brief Title: Presentation of Lumbar Disc and Reduction of Symptoms
Acronym: POLDAROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DT2656
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2008-05

CONDITIONS: Radiculopathy
Keywords: Intervertebral disc; Lumbar discectomy; Outcome; Radiculopathy due to prolapsed intervertebral disc.
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- experimental (Experimental): Participants are given their disc fragments following their operation
  Interventions: Behavioral: Presentation of excised intervertebral disc fragments

INTERVENTIONS:
Behavioral: Presentation of excised intervertebral disc fragments
  Arms: experimental

SUMMARY:
The trial aims to assess the hypothesis that presentation of the disc material to the patient following a lumbar microdiscectomy would positively influence the improvement in their leg and back symptoms.

DETAILED DESCRIPTION:
Objective. The trial aims to assess the hypothesis that presentation of removed material to the patient following a lumbar microdiscectomy would positively influence the improvement in their radiculopathic and degenerative symptoms.

Design. Data will be collected prospectively. Patient allocation to treatment groups will be by simple randomization using a computer generated sequence of random numbers. Trial participants will be blinded as to the trial hypothesis and investigators blinded to patient allocation.

Setting. Patients will all be treated in a single secondary care unit.

Participants. All adult patients undergoing a planned lumbar microdiscectomy for radiculopathy due to a prolapsed intervertebral disc over a six month period will be considered for entry into the trial. Exclusion criteria: inability to give verbal consent, age less than 18, previous spinal surgery, emergency discectomies, patients having spinal fusions and those with no radiculopathic symptoms.

Intervention. Patients allocated to the experimental arm will be given the removed disc fragments to keep once they have recovered from anaesthesia. Those in the control arm will not be shown disc fragments (best available treatment).

Main outcome measure. The degree of improvement in radiculopathic and degenerative symptoms reported by the patient at 2-3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing a planned lumbar microdiscectomy for radiculopathy due to a prolapsed intervertebral disc

Exclusion Criteria:

* inability to give verbal consent, age less than 18, previous spinal surgery, emergency discectomies, patients having spinal fusions and those with no radiculopathic symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Subjective experience of radiculopathic pain by the patient following surgery | 2-4 months

SECONDARY OUTCOMES:
Subjective experience of low back pain by the patient following surgery | 2-4 months
Subjective experience of lower limb motor weakness by the patient following surgery | 2-4 months
Subjective experience of paraesthesia by the patient following surgery | 2-4 months
Maximum walking distance | 2-4 months
Altered pattern of use of analgesia | 2-4 months
Subjective experience of numbness by the patient following surgery | 2-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Marios C Papadopoulos, DLitt, Principal Investigator — St George's, University of London
Locations (1):
- St George's Hospital, University of London, London, London, United Kingdom